CLINICAL TRIAL: NCT05146570
Title: Early Diagnosis and Treatment Monitoring of Native and Device-associated Meningitis Using D-lactate, a Pathogen-specific Diagnostic Biomarker in Cerebrospinal Fluid
Brief Title: Early Diagnosis of Native and Device-associated Meningitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andrej Trampuz, PD Dr. med, Head of Septic Surgery Unit, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DIAMEN
Record Dates: First submitted 2021-09-23; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Bacterial Meningitis; Fungal Meningitis; Implant Infection
Keywords: Pathogen-specific diagnostic biomarker; Cerebrospinal fluid; D-lactate; Device-associated meningitis; Diagnosis of meningitis
MeSH Terms: conditions — Meningitis, Bacterial; Meningitis, Fungal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aseptic Meningitis (Experimental): In all patients cerebrospinal (CSF) fluid will be aspirated following the routine diagnostic procedure. After aspiration CSF will be tested with standard diagnostic tests and experimental diagnostic test (D-lactate).
  Immediately after aspiration, 0.5-1 ml of cerebrospinal fluid will be transferred into each of the following vials:
  * native vial for conventional culture (agar plate & broth)
  * EDTA vial for the determination of leukocyte count and differential
  * pediatric blood culture bottle (BacTec PedsPlus/F)
  * native vial for biomarker detection (D-Lactate)
  Interventions: Diagnostic Test: D-lactate test; Diagnostic Test: Standard diagnostic tests
- Infective meningitis (Experimental): In all patients cerebrospinal (CSF) fluid will be aspirated following the routine diagnostic procedure. After aspiration CSF will be tested with standard diagnostic tests and experimental diagnostic test (D-lactate).
  Immediately after aspiration, 0.5-1 ml of cerebrospinal fluid will be transferred into each of the following vials:
  * native vial for conventional culture (agar plate & broth)
  * EDTA vial for the determination of leukocyte count and differential
  * pediatric blood culture bottle (BacTec PedsPlus/F)
  * native vial for biomarker detection (D-Lactate)
  Interventions: Diagnostic Test: D-lactate test; Diagnostic Test: Standard diagnostic tests

INTERVENTIONS:
Diagnostic Test: D-lactate test — In device-associated meningitis, CSF will be aspirated before, during or after surgery related to the device, according to the standard practice. Lumbar/ventricular punctures (pre-, intra- and/or postoperatively) and external ventricular (EVD) and lumbar drainage (ELD) aspiration will be performed by neurologist or neurosurgeon according to standardized aseptic techniques. In patients with native meningitis, CSF will be aspirated by lumbar puncture, according the standard practice. The D-lactate test will be performed using spectrophotometric enzyme assay according to the manufacturer's instructions (D-Lactate Colorimetric Assay).
Diagnostic Test: Standard diagnostic tests — In device-associated meningitis, CSF will be aspirated before, during or after surgery related to the device, according to the standard practice. Lumbar/ventricular punctures (pre-, intra- and/or postoperatively) and external ventricular (EVD) and lumbar drainage (ELD) aspiration will be performed by neurologist or neurosurgeon according to standardized aseptic techniques. In patients with native meningitis, CSF will be aspirated by lumbar puncture, according the standard practice. The standard diagnostic tests will be performed according to standard diagnostic laboratory instructions.

SUMMARY:
Device-associated meningitis is a severe complication after implantation of various central nervous system (CNS) devices such as ventriculoperitoneal (VP) and ventriculoatrial (VA) shunts, external ventricular drains (EVD), lumbar drains (ELD) and intrathecal pumps. In contrast to native meningitis, these infections are hard to diagnose both clinically and on the laboratory basis due to (i) atypical clinical manifestation, (ii) overlapping inflammation following surgery, and (iii) common culture negativity due to previous antibiotic therapy and slow growth of low-virulent pathogens. Also, device-associated infections are difficult to differentiate from aseptic shunt failure (dysfunction) or "chemical meningitis" caused by underlying neurosurgical condition that prompted the placement of the CNS device (e.g. intracranial hemorrhage).

Both native and device-associated meningitis carry substantial morbidity and mortality. Rapid and reliable diagnosis of meningitis is critical for initiating and choosing optimal treatment and minimizing the brain damage. Since treatment is different in septic than aseptic meningitis, it is paramount to diagnose or exclude septic meningitis as soon as possible.

Several new diagnostic methods, such as cerebrospinal fluid (CSF) procalcitonin, interleukin-6 and polymerase chain reaction (PCR) have been proposed for rapid diagnosis of meningitis. However, insufficient sensitivity and/or specificity, long time until test result, and complexity in handling or interpretation of results limit their use in clinical routine.

In previous studies CSF D-lactate test showed good specificity and sensitivity in patients with native meningitis. This biomarker is pathogen-specific - in contrast to other currently used host-specific biomarkers (leukocyte count, L-lactate, procalcitonin). However, no study on effectiveness of D-lactate test for the diagnosis of device-associated meningitis has been performed.

Successful management of device-associated meningitis depends upon appropriate control of the infectious complications. To deal with such complications, adequate assessment and prediction of the clinical course are needed. Another use of D-lactate test could be his role as prognostic factor of the clinical course of device-associated meningitis.

DETAILED DESCRIPTION:
Study aim Evaluation of the analytical and clinical performance (sensitivity, specificity, positive and negative predictive value, accuracy) of a novel, pathogen-specific biomarker D-lactate in the cerebrospinal fluid (CSF) for the diagnosis and treatment monitoring of native and device-associated meningitis. The performance of CSF D-lactate will be compared with currently used conventional CSF culture and biomarkers, using standard definition criteria for infection (native and device-associated meningitis).

Specific aims

* Aim 1. Determination of the performance of D-lactate test for the diagnosis of device-associated meningitis and native meningitis in serially collected CSF samples through lumbar/ventricular puncture (pre- or intra-operatively), external ventricular drainage (EVD), lumbar drainage (ELD) and shunt aspiration.
* Aim 2. Evaluate the optimal cut-off value of CSF D-lactate test for the diagnosis of device-associated and native meningitis using the existing definition criteria.
* Aim 3. Evaluation of performance of D-lactate test for the diagnosis of device-associated and native meningitis compared to standard tests (culture, gram stain, cerebrospinal fluid leukocyte count & differential, CSF lactate, CSF glucose, CSF-to-blood glucose ratio, CSF total protein, multiplex PCR) and novel biomarkers (CSF procalcitonin, alpha-defensin - ELISA, interleukin-6).

Study population:

Included will be consecutive patients with suspected device-associated meningitis and native meningitis treated in our institution. CSF will be aspirated following the routine diagnostic procedure. During conduction of this study no additional invasive or non-invasive examinations will be performed. The results obtained in this clinical investigation will not influence the diagnostic or treatment decisions for the patients.

Study definitions Device-associated meningitis will be defined according to modified criteria for nosocomial infections from Centers for Disease Control and Prevention (CDC).

Device-associated meningitis or ventriculitis must meet at least 1 of the following criteria:

1. Relevant growth of a pathogen in the CSF, on the device or in the wound swab of the device insertion site.
2. At least one of the following signs or symptoms without another identifiable cause: fever >38°C, headache, neck stiffness, cranial nerve signs, irritability, decrease in Glasgow coma scale (GCS) AND at least one of the following laboratory findings: increased CSF leukocytes (>5 × 10^6/l), increased CSF total protein (>0.45 g/l) or decreased CSF/blood glucose ratio (<0.5); positive CSF gram stain AND the physician initiates an antimicrobial therapy.

The following classification system for native meningitis will be applied:

Meningitis is diagnosed, if at least 1 of the following criteria is present:

1. Patient has organisms cultured from cerebrospinal fluid (CSF).
2. Patient has at least 1 of the following signs or symptoms: fever (>38°C), headache*, stiff neck*, meningeal signs*, cranial nerve signs*, or irritability*
3. And at least 1 of the following:

   1. increased white cells, elevated protein, and decreased glucose in CSF
   2. organisms seen on Gram's stain of CSF
   3. organisms cultured from blood
   4. positive laboratory test of CSF, blood, or urine
   5. diagnostic single antibody titer (IgM) or 4-fold increase in paired sera (IgG) for pathogen and if diagnosis is made antemortem, physician institutes appropriate antimicrobial therapy.

      * With no other recognized cause

In patients with diagnosed native or device-associated meningitis, the onset of the infection will be defined by clinical, laboratory and microbiology characteristics.

Study conduction In device-associated meningitis, CSF will be aspirated before, during or after surgery related to the device, according to the standard practice. Lumbar/ventricular punctures (pre-, intra- and/or postoperatively) and external ventricular (EVD) and lumbar drainage (ELD) aspiration will be performed by neurologist or neurosurgeon according to standardized aseptic techniques.

In patients with native meningitis, CSF will be aspirated by lumbar puncture, according the standard practice.

Laboratory procedure

* Immediately after aspiration, 0.5-1 ml of cerebrospinal fluid will be transferred into each of the following vials:

  * native vial for conventional culture (agar plate & broth)
  * EDTA vial for the determination of leukocyte count and differential
  * pediatric blood culture bottle (BacTec PedsPlus/F)
  * native vial for biomarker detection (e.g. D-Lactate, procalcitonin interleukin-6, alpha-defensin (ELISA) and additional tests (e.g. PCR)
* The D-lactate test will be performed using spectrophotometric enzyme assay according to the manufacturer's instructions (D-Lactate Colorimetric Assay. Sigma-Aldrich, St. Louis, Missouri, USA) as follows: the reaction mixture containing 10 µl of cerebrospinal fluid samples, 2 µl of substrate mix and 2 µl of enzyme mix and blank containing only the sample and substrate mix will be analyzed for each sample. A calibration curve with solutions of D-lactate (monolithium salt) in water will be processed in each batch. The mixture will be incubated at room temperature for 30 min and absorbance at 450 nm determined by Microplate Absorbance Reader. The optical density of each sample will be recalculated into D-lactate concentration in mmol.
* The test will be performed by two trained medical laboratory technical assistants, who are available during 12 hours on working days.
* All CSF aspirates and growing microorganisms (including those growing from intraoperative samples, such as peri-implant tissue or sonication fluid) will be stored in a biobank at -70°C. This fluid and culture collection allows subsequent additional analysis to assure the correct diagnosis.

Statistical analysis:

For device-associated meningitis it is assumed that 30-40% of the CSF samples are infected and the difference in sensitivity between D-lactate and conventional tests is 10% (90% for D-lactate vs. 80% for conventional tests). For native meningitis it is assumed that 10% of the CSF samples are infected and the difference in sensitivity between D-lactate and conventional tests is 20% (95% for D-lactate vs. 75% for conventional tests). Proof of non-inferiority between the two tests is provided by a one-sided two-group test of the percentage values. The non-inferiority is determined at a difference of 10% and can be shown for foreign material-associated meningitis in 458 patients and for native meningitis in 198 patients at a significance level of 5% and a power of 80%. The power calculation was performed with nQuery Advisor 7.0. Depending on the scale-type of data, the descriptive results are expressed as mean ± SD or number of subjects (percentage). Categorical variables will be compared using x2 or Fisher's exact tests, as appropriate. Continuous variables will be compared using the Wilcoxon rank-sum test. A p value <0.05 will be considered statistically significant. Test results will be evaluated with sensitivity, specificity, positive predictive value, negative predictive value, accuracy and statistical significance will be assessed with McNemar's Chi-squared test or a binomial test depending on sample size. All p-values from secondary analyses will be considered in a non-confirmatory exploratory manner. For statistical analyses the program packages SPSS (SPSS 10.0 for Windows, SPSS, USA) and the program package R (most recent version at time of analysis) will be used.

Investigators plan to include a total of 600 patients with device-associated meningitis and 220 patients with native meningitis. The high number of cases is indicated because investigators only expect a 30-40% infection rate for the foreign device-associated meningitis and a 10% infection rate for the native meningitis as well as a 10-15% drop-out rate (e.g. lack of leukocyte count or culture).

ELIGIBILITY:
Inclusion criteria:

* patients with suspected (clinical, paraclinical or radiological) native or device-associated meningitis
* age >18 years
* patient signs written consent to participate in the study

Exclusion criteria:

* inability of the patient or family member to consent to the study
* time from puncture to laboratory evaluation> 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 842 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Performance of D-lactate test for the diagnosis of native and device-associated meningitis. | up to 30 months
  Determined performance (D-lactate cut-off value, sensitivity, specificity, positive predictive value, negative predictive value, positive likelihood ratio, negative likelihood ratio) of D-lactate test.
  * The Mann-Whitney test and Spearman's correlation will be applied to analyze the quantitative variables. Youden's J statistic will be used for determining optimal D-lactate cut-off value on the receiver operating characteristic (ROC) curve by maximizing sensitivity and specificity.
  * The area under the ROC curves will be calculated to compare the D-lactate test performance.

SECONDARY OUTCOMES:
Performance of the D-lactate test in comparison with standard tests for the diagnosis of native and device-associated meningitis. | up to 30 months
  Identified differences between performance of D-lactate test and standard tests (cultures, cell counting, Gram preparations, L-lactate, protein and glucose) for the diagnosis of native and device-associated meningitis.
  - To compare the performances of different tests (sensitivity, specificity, positive predictive value, negative predictive value, positive likelihood ratio, negative likelihood ratio) the McNemar chi-square will be used.
Treatment monitoring using D-lactate test (as a predictor of treatment success / failure). | up to 30 months
  Number of participants with cured (or recurrent) native and device-associated meningitis assed by D-lactate test and with standard diagnostic criteria.
  * D-lactate test will be judged positive or negative according to the established cut-off in Outcome 1.
  * Standard methods include standard diagnostic criteria for device-associated meningitis according to modified criteria for nosocomial infections from Centers for Disease Control and Prevention (CDC) and standard diagnostic criteria for native meningitis (according to study description).

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Trampuz, PD Dr. med, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hasbun R. Central Nervous System Device Infections. Curr Infect Dis Rep. 2016 Nov;18(11):34. doi: 10.1007/s11908-016-0541-x. PMID 27686676
- [Background] van de Beek D, Drake JM, Tunkel AR. Nosocomial bacterial meningitis. N Engl J Med. 2010 Jan 14;362(2):146-54. doi: 10.1056/NEJMra0804573. No abstract available. PMID 20071704
- [Background] Conen A, Walti LN, Merlo A, Fluckiger U, Battegay M, Trampuz A. Characteristics and treatment outcome of cerebrospinal fluid shunt-associated infections in adults: a retrospective analysis over an 11-year period. Clin Infect Dis. 2008 Jul 1;47(1):73-82. doi: 10.1086/588298. PMID 18484878
- [Background] Banks JT, Bharara S, Tubbs RS, Wolff CL, Gillespie GY, Markert JM, Blount JP. Polymerase chain reaction for the rapid detection of cerebrospinal fluid shunt or ventriculostomy infections. Neurosurgery. 2005 Dec;57(6):1237-43; discussion 1237-43. doi: 10.1227/01.neu.0000186038.98817.72. PMID 16331172
- [Background] Li Y, Zhang G, Ma R, Du Y, Zhang L, Li F, Fang F, Lv H, Wang Q, Zhang Y, Kang X. The diagnostic value of cerebrospinal fluids procalcitonin and lactate for the differential diagnosis of post-neurosurgical bacterial meningitis and aseptic meningitis. Clin Biochem. 2015 Jan;48(1-2):50-4. doi: 10.1016/j.clinbiochem.2014.10.007. Epub 2014 Oct 30. PMID 25445228
- [Background] Chen Z, Wang Y, Zeng A, Chen L, Wu R, Chen B, Chen M, Bo J, Zhang H, Peng Q, Lu J, Meng QH. The clinical diagnostic significance of cerebrospinal fluid D-lactate for bacterial meningitis. Clin Chim Acta. 2012 Oct 9;413(19-20):1512-5. doi: 10.1016/j.cca.2012.06.018. Epub 2012 Jun 17. PMID 22713513
- [Background] Walti LN, Conen A, Coward J, Jost GF, Trampuz A. Characteristics of infections associated with external ventricular drains of cerebrospinal fluid. J Infect. 2013 May;66(5):424-31. doi: 10.1016/j.jinf.2012.12.010. Epub 2013 Jan 9. PMID 23313468
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699